CLINICAL TRIAL: NCT03198312
Title: a Prospective, Multicenter, Randomized, Open, Parallel Controlled Noninferiority Clinical Study to Evaluate the Efficacy and Safety of CathiportTM Implantable Drug Delivery Device
Brief Title: CathiportTM Clinical Efficacy and Safety Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Branden-abc
Record Dates: First submitted 2017-05-25; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CathiportTM (Experimental): be used for all kinds of high concentrations of chemotherapeutic drugs, completely parenteral nutrient solution infusion, blood transfusion and blood samples.
  Interventions: Device: CathiportTM
- Implant Port (Active Comparator): be used for all kinds of high concentrations of chemotherapeutic drugs, completely parenteral nutrient solution infusion, blood transfusion and blood samples.
  Interventions: Device: Implant Port

INTERVENTIONS:
Device: CathiportTM — fully implanted
  Arms: CathiportTM
Device: Implant Port — fully implanted
  Arms: Implant Port

SUMMARY:
Develop a prospective, multicenter, randomized, open, parallel controlled noninferiority clinical trial to evaluate the efficacy and safety of CathiportTM implantable drug delivery device

DETAILED DESCRIPTION:
I-Port is also called the implantable infusion Port typed central venous catheter and suite, it is a kind of the closed venous infusion system that can fully implanted, can be used for all kinds of high concentrations of chemotherapeutic drugs, completely parenteral nutrient solution infusion, blood transfusion and blood samples, It can be used to reduce painfulness and the difficulty of repeated venipuncture, to prevent external stimulants weeks vein injury, and the daily life of patients is not limited, they don't need to change medicine, can bathe, so can improve the quality of life.

The purpose of the study is to evaluate the safety and efficacy of the CathiportTM. The CathiportTM will be compared to an active control group represented by the FDA approved commercially available Bard Implant Port.

The study consists of a randomized clinical trial (RCT) in China which will enroll approximately 220 subjects (1:1 randomization CathiportTM : Implant Port) with patients required repeated and chronic drug input and fluid.

All subjects in the RCT will be screened per the protocol required inclusion/exclusion criteria. The data collected will be compared to data from the subjects enrolled into the Implant Port of US RCT.

All subjects will have clinical follow-up at 1, 2, 3, 4, 5, 6 months and be provided nursing service to t maintain he Port , and verify whether the pipe is blocked and to prevent the Port into the liquid pipe clogging, and to observe the hematoma and infection situation of the operation or puncture points, observe whether if there is blocking pipe, and fluid extravasation surrounding skin tissue of judging when using, whether there are conditions such as shift or discount.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old;
2. Need for long-term intravenous fluids;
3. Lack of peripheral venous access ;
4. Need stimulants infusion, such as chemotherapy drugs;
5. Need infusion of high permeability or sticky liquid, such as parenteral nutrient solution, fat emulsion;
6. Need repeated blood or blood products transfusion and repeated blood collection;
7. Fit and need implanted Port;
8. Willing to participate in clinical research and signed informed consent;

Patient meet 1 and 8 firstly, and then meet any one item with 2-7 above can be accepted.

Exclusion Criteria:

1. Cancer patients whose vascular related to the surgery is compressed ;
2. Women patients with pregnancy and lactation;
3. Participate other studies before achieving the primary end point already;
4. Confirmed or suspected catheter-related infections, disseminated intravascular coagulation, bacteremia, sepsis;
5. Body size is not suitable for implanting the infusion port ;
6. Confirmed or suspected allergic to silicone material;
7. Having a history of radiation therapy at the pre-implant site;
8. Having occurred acute myocardial infarction within 1 week or stroke in the past 6 months;
9. Having a history of venous thrombosis, trauma, or vascular surgery;
10. Superior vena cava syndrome;
11. Having poor compliance behavior;
12. Having installed the cardiac pacemaker device, bypass, accepted heart transplant or diagnosed with kidney failure（GFR≤30ml/Min）.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-10-20 (Estimated); Study Completion 2018-01-20 (Estimated)

PRIMARY OUTCOMES:
Normal usage rate of the equipment | at 6 months
  The probability of normally drugs or liquid infusion

SECONDARY OUTCOMES:
Success rate of equipment | 0 to 24 hours after implantation
  Refers to the equipment can be get to the therapeutic part as expected successfully , the catheter can infused smoothly and the blood samples can be get back normally
Success rate of surgery | 0 to 24 hours after operation
  The fluid can be infused and withdraw normally, and no pneumothorax, air embolism, mediastinal hematoma surgical complications appeared
the evaluation of the efficiency | at 1,2,3,4,5,6 month
  Catheter indwelling time
the evaluation of the convenience | intraoperative
  all the operaters will give a convenience evaluation timely by answering the questionnare
the evaluation of the comfort | intraoperative
  physical performance evaluation of the device